CLINICAL TRIAL: NCT01716858
Title: Sulforaphane-rich Broccoli Sprout Extract for Schizophrenia
Brief Title: An Open Study of Sulforaphane-rich Broccoli Sprout Extract in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Kenji Hashimoto, Sulforaphane for Schizophrenia, Chiba University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chiba_SFN_Openstudy2012
Record Dates: First submitted 2012-10-22; First posted 2012-10-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2012-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Sulforaphane; Psychosis; Cognition; Oxidative stress; Antioxidant; Anti-inflammatory
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A single-arm study (Experimental)
  Interventions: Dietary Supplement: Sulforaphane-rich Broccoli Sprout Extract

INTERVENTIONS:
Dietary Supplement: Sulforaphane-rich Broccoli Sprout Extract

SUMMARY:
Accumulating evidence suggests a role of oxidative stress in the pathophysiology of schizophrenia. The potent antioxidant sulforaphane (SFN) is an organosulfur compound derived from a glucosinolate precursor found in cruciferous vegetables such as broccoli, Brussels sprouts and cabbage. The protection afforded by SFN is thought to be mediated via activation of the NF-E2-related factor-2 (Nrf2) pathway and subsequent up-regulation of phase II detoxification enzymes and antioxidant proteins, through an enhancer sequence referred to as the electrophilic responsive element or antioxidant responsive element. Recently, we reported that SFN could attenuate behavioral abnormalities in mice after the NMDA receptor antagonist phencyclidine. Considering the potent antioxidant effects of SFN, we have a hypothesis that SFN would be a potential therapeutic drug for schizophrenia. The purpose of this study is to determine whether SFN-rich broccoli sprout extract have beneficial effects in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia for DSM-IV TR criteria
* Patients are treated with an antipsychotic drug (risperidone, olanzapine, quetiapine, perospirone, aripiprazole, blonanserin, paliperidone).
* Patients are stable for 4-weeks for antipsychotic medication.

Exclusion Criteria:

* Patients treated with clozapine
* Patients treated with two or more antipsychotic drugs
* Pregnant or breast-feeding women
* Patients treated with sulforaphane for more than 8-weeks in the past.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Change from baseline in PANSS scores at 8-weeks

SECONDARY OUTCOMES:
Cognition using CogState Research Battery | Change from baseline in the scores of the battery at 8-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masaomi Iyo, MD, PhD, Study Chair — Chairman, Department of Psychiatry, Chiba University Graduate School of Medicine
Locations (1):
- Chiba University Hospital, Chiba, Chiba, Japan

REFERENCES:
- [Result] Shiina A, Kanahara N, Sasaki T, Oda Y, Hashimoto T, Hasegawa T, Yoshida T, Iyo M, Hashimoto K. An Open Study of Sulforaphane-rich Broccoli Sprout Extract in Patients with Schizophrenia. Clin Psychopharmacol Neurosci. 2015 Apr 30;13(1):62-7. doi: 10.9758/cpn.2015.13.1.62. PMID 25912539
- See also: Related Info — http://www.cpn.or.kr/journal/view.html?volume=13&number=1&spage=62